CLINICAL TRIAL: NCT01676298
Title: Study of the Analytical Reproducibility of the Spartan FRX CYP2C19 *2,*3 and *17 Genotyping System.
Brief Title: Spartan FRX Project Reproducibility Study
Status: Completed | Type: Observational
Sponsor: Spartan Bioscience Inc. (Industry)
Collaborators: Children's Hospital of Eastern Ontario (Other); Ottawa Hospital Research Institute (Other); Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 01001686
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-12

CONDITIONS: Analytical Reproducibility of a Medical Device
Keywords: Cyp2C19; Genotyping; Spartan; Reproducibility

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Spartan FRX CYP2C19 Test System

SUMMARY:
The Spartan FRX CYP2C19 Test System (hereafter referred to as the 'FRX System') is a qualitative in vitro diagnostic test for the identification of a patient's CYP2C19 *2, *3 and *17 genotypes from genomic DNA obtained from buccal swab samples. The objective of the study is to evaluate the performance of the FRX System under multivariate conditions including different days, sites, operators and systems.

DETAILED DESCRIPTION:
The FRX system is comprised of hardware and consumable components. The hardware components of the system include an Analyzer (thermal cycler with fluorescence detection capability), a notebook computer and a printer. The consumable component of the FRX system is a sample collection kit. Each kit contains a buccal swab (used to collect the patient sample) and a tube containing the reagents required for genomic DNA extraction and PCR (polymerase chain reaction) amplification stages of the test.

The Spartan FRX System is capable of detecting three CYP2C19 SNPs(single nucleotide polymorphism) (*2, *3, *17) in each test performed. An individual sample collection kit is required for each SNP tested; therefore three sample collection kits are required for each test performed on the system.

To perform a test, the user collects three buccal samples from the patient and then inserts a sample into each of the three reagent tubes (one for each of the CYP2C19 loci *2, *3 and *17). The reagent tubes are placed into the Analyzer and the FRX system automates the processes of DNA extraction, PCR amplification, fluorescent signal detection and data analysis. The system provides the user with a printed result listing the patient genotypes at the *2, *3 and *17 loci.

The objective of the study is to evaluate the performance of the FRX System under multivariate conditions. Specifically, the following variables will be included in the study:

* Test site - x3
* Operator - x6 (2 per site)
* Day - x15 (5 non-consecutive days per site)
* FRX System - x16

Test performance is defined as the number of correct genotype calls, expressed as a percentage of the total number of tests performed on the system.

For both the first-pass and second-pass results, 1-sided 95% confidence lower limits will be calculated using the score method for the % correct calls (i.e. % agreement).

Genotype results from the FRX system will be compared with results of DNA sequencing. The result of the FRX System test will be determined to be correct if the genotype calls for all three SNPs are identical to the genotypes determined by DNA sequencing for that sample/individual.

Results of the Reproducibility Study will be acceptable if the lower bound of a 1-sided 95% confidence limit of the total correct call rate per genotype is greater than or equal to 95%, based on second-pass results.

ELIGIBILITY:
Inclusion Criteria:

* Above 16 years of age
* Must have required genotype

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 8 Individuals with predetermined CYP2C19 *2,*3 and *17 genotypes
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris JE Harder, PhD, Principal Investigator — Spartan Bioscience; Azar Azad, PhD, Principal Investigator — MOUNT SINAI HOSPITAL; Marc Desjardins, PhD, Principal Investigator — Ottawa Hosptial Research Institute; Jean McGowan-Jordan, PhD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (3):
- Canada (3):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Mount Sinai Services, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 individuals were recruited for a company pool of known suspected genotypes; each with a different CYP2C19 genotype confirmed prior to the study by bi-directional sequencing.
Pre-assignment Details: Spartan Bioscience
Groups:
- *1/*1 CYP2C19 Genotype; *1/*2 CYP2C19 Genotype; *2/*2 CYP2C19 Genotype; *3/*1 CYP2C19 Genotype; *1/*17 CYP2C19 Genotype; *17/*17 CYP2C19 Genotype; *2/*3 CYP2C19 Genotype; *2/*17 CYP2C19 Genotype: Subject had genotype confirmed via bi-directional sequencing.
Period: Overall Study
Arm/Group | *1/*1 CYP2C19 Genotype | *1/*2 CYP2C19 Genotype | *2/*2 CYP2C19 Genotype | *3/*1 CYP2C19 Genotype | *1/*17 CYP2C19 Genotype | *17/*17 CYP2C19 Genotype | *2/*3 CYP2C19 Genotype | *2/*17 CYP2C19 Genotype
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
All Genotypes Confirmed With Reference | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Participated in All Tests | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | *1/*1 CYP2C19 Genotype | *1/*2 CYP2C19 Genotype | *2/*2 CYP2C19 Genotype | *3/*1 CYP2C19 Genotype | *1/*17 CYP2C19 Genotype | *17/*17 CYP2C19 Genotype | *2/*3 CYP2C19 Genotype | *2/*17 CYP2C19 Genotype | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 7
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3
  Male | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Correct Calls to Assess Reproducibility of the Spartan FRX CYP2C19 System.
Description: Reproducibility was calculated as a percentage of the correct calls over the total calls made for each genotype group. All calls were made using the Spartan FRX CYP2C19 genotyping diagnostic system.
  All data analyses was qualitative, based on the genotype calls determined by the FRX system (using on-board automated data analysis). A printed result listing the genotype call for each SNP was generated by the FRX system at the end of each run. If the result of a test is "Inconclusive" for one or more SNPs, the test were immediately repeated for the corresponding SNP(s) only, per the instructions for use. Results are reported based on both first-pass and second-pass (i.e. repeated test). For both the first-pass and second-pass results, 1-sided 95% confidence lower limits were calculated using the score method for the % correct calls (i.e. % agreement).
Time Frame: After second pass result is complete (~3h)
Measure: Number (95% Confidence Interval); unit: Percentage of Correct Calls
Units Other Than Participants: CYP2C19 Genotype
Arm/Group | *1/*1 CYP2C19 Genotype | *1/*2 CYP2C19 Genotype | *2/*2 CYP2C19 Genotype | *3/*1 CYP2C19 Genotype | *1/*17 CYP2C19 Genotype | *17/*17 CYP2C19 Genotype | *2/*3 CYP2C19 Genotype | *2/*17 CYP2C19 Genotype
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Number analyzed (CYP2C19 Genotype) | 120 | 120 | 200 | 120 | 120 | 120 | 120 | 120
Percentage of Correct Calls | 98.3 [95.1 to 99.4] | 100 [97.8 to 100] | 97.5 [95 to 98.8] | 99.2 [96.4 to 99.8] | 100 [97.8 to 100] | 99.2 [96.4 to 99.8] | 99.2 [96.4 to 99.8] | 99.2 [96.4 to 99.8]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the full duration of the trial (~2 months).
Description: No adverse events were encountered.
Arm/Group | *1/*1 CYP2C19 Genotype | *1/*2 CYP2C19 Genotype | *2/*2 CYP2C19 Genotype | *3/*1 CYP2C19 Genotype | *1/*17 CYP2C19 Genotype | *17/*17 CYP2C19 Genotype | *2/*3 CYP2C19 Genotype | *2/*17 CYP2C19 Genotype
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less